CLINICAL TRIAL: NCT01079078
Title: An Open Label, Balanced, Randomised, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioavailability Study Comparing Acetaminophen 650 mg Extended Release Gelcaps (Containing Acetaminophen 650 mg) of OHM Laboratories (A Subsidiary of Ranbaxy Pharmaceuticals Inc.) With TylenolÒ Arthritis Pain Extended Release Caplets (Containing Acetaminophen 650 mg) of McNeil-PPC Inc. in Healthy, Adult, Human, Male Subjects Under Fed Condition.
Brief Title: A Relative Bioavailability Study of Acetaminophen 650 mg Extended Release Gelcaps Under Fed Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 144_ACETA_07
Record Dates: First submitted 2010-02-18; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Acetaminophen fed study
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Acetaminophen extended release gelcaps 650 mg of OHM Laboratories Inc. (a subsidiary of Ranbaxy Pharmaceuticals Inc.)
  Interventions: Drug: Acetaminophen
- Reference (Active Comparator): Tylenol® Arthritis Pain caplets 650 mg (containing acetaminophen 650 mg)of McNeil Consumer & Specialty Pharmaceuticals, Division of MCNEIL-PPC, Inc. Fort Washington, PA 19034 USA
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen

SUMMARY:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single dose, crossover bioavailability study comparing acetaminophen extended release gelcaps 650 mg (containing acetaminophen 650 mg) of OHM Laboratories Inc. with TYLENOLÒ arthritis pain caplets 650 mg (containing acetaminophen 650 mg) of McNeil Consumer & specialty Pharmaceuticals in healthy, adult, human, male subjects under fed condition.

DETAILED DESCRIPTION:
A single oral dose of acetaminophen 650 mg was administered (except Subject No. 17) with 240 mL of drinking water during each period under supervision of trained study personnel.

During the course of the study, safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical, serology parameters and urine analysis) at base line. Laboratory parameters of hematology and biochemistry were repeated at the end of study (except Glucose and cholesterol).

ELIGIBILITY:
Inclusion Criteria:

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for the corresponding height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.
* Were non-vegetarian.

There was no deviation in this regard.

Exclusion Criteria:

* Had a history of hypersensitivity to acetaminophen or to any of the components of the formulation.
* Had a history of skin rashes, thrombocytopenia, urticaria or angioedema.
* Had a history of peptic ulcer.
* Had recent history of nausea and vomiting
* Showed any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Showed presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Showed presence of values which were significantly different from normal reference ranges defined and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Were positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Showed presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Showed clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) or protein (positive).
* Showed clinically abnormal ECG or Chest X-ray.
* Had a history of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
* Had a history of any psychiatric illness, which might impair the ability to provide written informed consent.
* Were regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
* Had history of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

There was no deviation in this regard.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of acetaminophen 650 mg extended release gelcaps under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Unit, Majeedia Hospital (2nd Floor), New Delhi, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html